CLINICAL TRIAL: NCT05543733
Title: Home Exercise And Resiliency Training (HEART) Club: A Virtual Care at Home Program to Reduce Frailty for Adults With Fontan Circulation
Brief Title: Home Exercise And Resiliency Training (Heart) Club
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jesse Hansen, Assistant Professor of Pediatrics, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00220044
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fontan Physiology; Frailty
Keywords: Exercise program; Liver stiffness
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home exercise program (Experimental)
  Interventions: Behavioral: Home exercise program

INTERVENTIONS:
Behavioral: Home exercise program — Participants will complete a 6-month prescription telemedicine-based structured home exercise program. Baseline information will be used to develop a personalized home exercise program. This program will involve downloading the MyDataHelps application on a mobile device to securely collect wearable device information like step counts, activity minutes, and heart rate. Additionally, participants will have multiple virtual visits as well as the 2 in-person visits.

SUMMARY:
The purpose of this research study is to evaluate the impact of a telemedicine-based structured home exercise program on frailty and exercise capacity in individuals with Fontan heart physiology, demonstrate that a telemedicine exercise program reduces socioeconomic and geographic barriers to access to exercise training, and to explore the impact of a structured exercise program on markers of Fontan-associated liver disease.

DETAILED DESCRIPTION:
This study will require two in-person visits to the exercise physiology lab as well as virtual follow-up visits. Visit one will require participants to complete a cardiopulmonary exercise test (CPET), liver ultrasound, 6-minute walk, grip strength test, arm circumference measure, body composition analysis, anthropometrics measurement, surveys and a biomarker blood sample collection. The second in-person visit will require participants to complete a final cardiopulmonary exercise test, liver ultrasound, 6-minute walk, grip strength test and arm circumference, biomarker blood sample and final survey.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with Fontan physiology
* 19 years old at age of enrollment

Exclusion Criteria:

* Height less than 130 centimeter (cm)
* Pregnancy or the plan to become pregnant during the study period
* Current intravenous inotropic drugs
* Severe ventricular dysfunction assessed qualitatively by clinical echocardiography within six months prior to enrollment
* Severe valvar regurgitation, ventricular outflow obstruction, or aortic arch obstruction assessed by clinical echocardiography within six months prior to enrollment
* History of arrhythmia with exercise (excluding isolated supraventricular or ventricular ectopy without symptoms)
* Inability to complete exercise testing at baseline screening
* Noncardiac medical, psychiatric, and/or social disorder that would prevent successful completion of planned study testing or would invalidate its results

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Frailty score by the Fried frailty instrument | day 1 (baseline), week 26 (final visit)
  The questionnaire evaluates five components of the frailty syndrome (weakness, slowness, shrinkage, exhaustion, and diminished physical activity). Sum of the components will have a possible score of 0-5: not frail (score 0), pre-frail (score 1-2), frail (score great or equal to 3), undetermined (missing component).

SECONDARY OUTCOMES:
Change in 7-day average step count over 6 month period | Baseline, 6 months
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) - 29 | day 1 (baseline), week 26 (final visit)
  This survey has 29 items across the following domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, ability to participate in social roles and activities, cognitive function on a scale of 1 (worst) to 5 (best), and pain intensity (on a scale ranging from 0 (no pain) to 10 (worst pain imaginable).
Change in 6-minute walk distance | day 1 (baseline), week 26 (final visit)
Change in peak oxygen consumption | day 1 (baseline), week 26 (final visit)
  This is measured during a Cardiopulmonary Exercise Testing (CPET) test measured in milliliters per minute (mL/min).
Change in oxygen consumption at anaerobic threshold | day 1 (baseline), week 26 (final visit)
  This is measured during a CPET.
Change in liver stiffness measured by ultrasound | day 1 (baseline), week 26 (final visit)
  This is measured during ultrasound, units meters per second (m/sec)
Change in alpha fetoprotein (AFP) | day 1 (baseline), week 26 (final visit)
  This is a blood sample.
Change in Aspartate Transferase (AST) | day 1 (baseline), week 26 (final visit)
  This is a blood sample.
Change in Alanine Aminotransferase (ALT) | day 1 (baseline), week 26 (final visit)
  This is a blood sample.
Change in platelets | day 1 (baseline), week 26 (final visit)
  This is a blood sample.
Change in Gamma-glutamyl Transferase (GGT) | day 1 (baseline), week 26 (final visit)
  This is a blood sample.
Change in Enhanced Liver Fibrosis (Elf) Score number | day 1 (baseline), week 26 (final visit)
  This is a blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hansen, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No